CLINICAL TRIAL: NCT06720870
Title: An Italian Multicenter Retrospective Observational Study to Assess Effectiveness and Safety of Siltuximab for Patients with Castleman's Disease Treated in Italy in a Real-life Context
Acronym: SilOs
Status: Recruiting | Type: Observational
Sponsor: IRCCS Azienda Ospedaliero-Universitaria di Bologna (Other)
Responsible Party: Sponsor
Other Study IDs: SilOs
Record Dates: First submitted 2024-12-03; First posted 2024-12-06 (Actual); Last update posted 2024-12-06 (Actual); Status verified 2024-10

CONDITIONS: Castleman Disease
Keywords: Siltuximab
MeSH Terms: conditions — Castleman Disease

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Retrospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

SUMMARY:
The study is a pilot, observational, retrospective, and (italian) multicenter study.

The study will involve the collection of patient data from medical records for patients with Multicentric Castelman Disease Relapsed/Refractory who received treatment with at least one dose of siltuximab, as part of standard of care in a real-life context, from July 2016 till April 2022 in 31selected italian centres.

DETAILED DESCRIPTION:
The aim of the present study is to provide useful information about use, effectiveness, and safety profile of siltuximab given to relapsed or refractory (R/R) MCD in a real-life context since approval as more data are needed to improve knowledge in this rare disease. The observational, non-interventional nature of the study is based on the retrospective observation of current clinical practice without the application of any kind of ad hoc 'intervention' for the study itself. Infact, patients participating in the study will not be subjected to any procedures outside the normal clinical practice; likewise, the clinical variables that will be collected for the study are those that are already commonly collected by the physicians in clinical practice.

ELIGIBILITY:
Inclusion Criteria:

1. Histologically confirmed diagnosis of R/R MCD HIV and HHV-8 negative patients who underwent siltuximab in a real-life context from July 2016 till April 2022.
2. Age ≥ 18 yearsatenrollment
3. Signature of written informed consent (where applicable)

Exclusion Criteria:

1. R/R MCD patients who underwent siltuximab in a clinical trial context

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Patients with R/R MCD who receive at least one dose of siltuximab in a real-life context from July 2016 till April 2022.
Sampling Method: Non-Probability Sample
Enrollment: 65 (Estimated)
Dates: Start 2023-03-01 (Actual); Primary Completion 2025-01 (Estimated); Study Completion 2025-01 (Estimated)

PRIMARY OUTCOMES:
overall response rate (ORR) | after the end of siltuximab infusion
  Primarily this study aims to evaluate retrospectively effectiveness in terms of ORR of siltuximab as a single agent in patients with R/R MCD treated with at least one dose of siltuximab in a real-life context

SECONDARY OUTCOMES:
Duration of response (DoR) | before, during and after the end of siltuximab infusion
  Duration of response (DoR)
Progression-free survival (PFS) | before, during and after the end of siltuximab infusion
  Progression-free survival (PFS)
Overall Survival (OS) | before, during and after the end of siltuximab infusion
  Overall Survival (OS)
Duration Free Survival (DFS) | before, during and after the end of siltuximab infusion
  Duration Free Survival (DFS)
Best response rate (BRR) | before, during and after the end of siltuximab infusion
  Best response rate (BRR)
safety and tolerability of siltuximab | before, during and after the end of siltuximab infusion
  safety and tolerability of siltuximab

CONTACTS AND LOCATIONS:
Overall Officials: Pier Luigi Zinzani, MD, Principal Investigator — IRCCS Azienda Ospedaliero-Universitaria di Bologna
Locations (12):
- Italy (12):
  - IRCCS Azienda Ospedaliero - Universitaria di Bologna, Bologna, Bologna
  - Azienda Ospedaliera Sant'Anna e San Sebastiano, Caserta, Caserta
  - Policlinico di Bari - Azienda Ospedaliero Universitaria Consorziale Policlinico, Bari
  - Azienda Ospedaliera Universitaria Arcispedale Sant'Anna, Ferrara
  - Azienda Ospedaliero Universitaria Careggi, Florence
  - Irccs Ospedale San Raffaele, Milan
  - Azienda Ospedaliero-Universitaria "Maggiore della Carità", Novara
  - Azienda Ospedaliera Di Padova, Padua
  - Fondazione IRCCS Policlinico San Matteo, Pavia
  - Azienda Ospedaliera Universitaria Senese, Siena
  - Azienda ULSS 2 Marca Trevigiana - UOC Medicina Interna 1 Centro di Riferimento per le Malattie Rare del Sistema Immunitario e dell'Apparato Respiratorio, Treviso
  - Azienda Ulss 2 Marca Trevigiana- Ospedale Di Treviso, Treviso

IPD SHARING:
Plan to Share IPD: No